CLINICAL TRIAL: NCT07402824
Title: Investigation of Mobbing Exposure and Job Satisfaction Levels Among Physiotherapists
Brief Title: Mobbing Exposure and Job Satisfaction Among Physiotherapists
Status: Recruiting | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ismail Okur, Assst. Prof., Kutahya Health Sciences University
Other Study IDs: KHSU- 2025/04-25
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Job Satisfaction; Bullying, Workplace
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physical Therapists: Having graduated from at least a 4-year undergraduate program in Physiotherapy and Rehabilitation.

SUMMARY:
Physiotherapists, who hold a significant place in the healthcare sector, are at risk for mobbing and low levels of job satisfaction due to both demanding physical working conditions and emotional stress. This study was designed to investigate the mobbing exposure and job satisfaction levels of physiotherapists.

ELIGIBILITY:
Inclusion Criteria:

* Currently working or having previously worked as a physiotherapist in Turkey.
* Graduation from a minimum 4-year Physiotherapy and Rehabilitation degree program.
* Voluntary participation.

Exclusion Criteria:

* Forms with incorrect answers to dummy questions (trap questions).
* Forms with missing data.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of physiotherapists who are currently practicing or have previously practiced in Turkey. The participants include professionals who have completed at least a 4-year undergraduate degree in Physiotherapy and Rehabilitation. This population encompasses individuals working across various healthcare settings (e.g., public hospitals, private clinics, rehabilitation centers) to provide a comprehensive understanding of the relationship between mobbing exposure and job satisfaction levels within the profession.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02-04 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Mobbing Scale Description | Baseline
  The Mobbing Scale was developed by Aiello et al. (2008) to measure the perception of workplace bullying. The Turkish validity and reliability study was conducted by Laleoğlu and Özmete (2013), with a Cronbach's Alpha coefficient of 0.94. The scale consists of 38 items rated on a 7-point Likert-type scale.
Minnesota Job Satisfaction Questionnaire (MSQ) - Short Form Description: | Baseline
  The MSQ was developed by Weiss et al. (1967) to evaluate job satisfaction, and the Turkish validity and reliability study was performed by Baycan (1985). It is a 20-item, 5-point Likert-type scale. Each item is scored from 1 to 5. Total Score Range: 20 to 100. Higher scores indicate higher levels of job satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Kütahya, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Szczegielniak A, Skowronek A, Krysta K, Krupka-Matuszczyk I. Aggression in the work environment of physiotherapists. Psychiatr Danub. 2012 Sep;24 Suppl 1:S147-52. PMID 22945210